Using fMRI and sEMG to Evaluate the Effects and Mechanism on Abdominal Acupuncture Combined With Upper Limb Rehabilitation Training on Brain Plasticity of Hemiplegic Patients With Stroke

Head of Clinical Research Unit: Guangdong Provincial Hospital of

Chinese Medicine

**Director of Clinical Research:** Chen Hongxia

Clinical Research Participating Unit: Guangdong Provincial Hospital of

Chinese Medicine ,Chinese

University of Hong Kong .

Reporting Unit: Guangdong Provincial Hospital of Chinese Medicine

Research Director: Chen Hongxia

## **Statistical Analysis Plan**

Statistical analysis of our research will use SPSS 18.0 and MATLAB statistical software. The measurement data adopt T-Test, counting data use repeated measurement variance analysis and X2 test. And the image analysis adopt SPM8 software.